CLINICAL TRIAL: NCT04762810
Title: A Prospective Study to Evaluate the Efficacy and Safety of Cyclophosphamide in the Treatment of Idiopathic Retroperitoneal Fibrosis
Brief Title: A Prospective Study of Cyclophosphamide Treatment for Idiopathic Retroperitoneal Fibrosis
Acronym: IRPF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cyclophosphamide for IRPF
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Retroperitoneal Fibrosis
MeSH Terms: conditions — Retroperitoneal Fibrosis | interventions — Cyclophosphamide; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclophosphamide and Glucocorticoids (Experimental): Through the selective depletion of proliferating lymphocytes, cyclophosphamide has an inhibitory effect on both humoral and cellular immunity. Cyclophosphamide 50mg per day for 6 months and decrease to 50mg Qod for 6 months.
  Interventions: Drug: Cyclophosphamide and glucocorticoids
- Glucocorticoids monotherapy (Active Comparator): Prednisone/prednisolone: started at 0.6-0. 8mg/kg.d for 2 to 4 weeks, tapered at 5mg per 1-2 weeks before 15mg per day, and tapered at 2.5-5mg per 2 weeks to equal to or less than 5mg per day in 6 months.
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: Cyclophosphamide and glucocorticoids — Prednisone/prednisolone: started at 0.6-0. 8mg/kg.d for 2 to 4 weeks, tapered at 5mg per 1-2 weeks before 15mg per day, and tapered at 2.5-5mg per 2 weeks to equal to or less than 5mg per day in 6 months. Cyclophosphamide 50mg per day for 6 months and decrease to 50mg Qod for 6 months.
  Arms: Cyclophosphamide and Glucocorticoids
Drug: Glucocorticoids — Steroids have fast onset of action and multiple anti-inflammatory effects. Prednisone/prednisolone: started at 0.6-0. 8mg/kg.d for 2 to 4 weeks, tapered at 5mg per 1-2 weeks before 15mg per day, and tapered at 2.5-5mg per 2 weeks to equal to or less than 5mg per day in 6 months.
  Arms: Glucocorticoids monotherapy

SUMMARY:
This prospective, interventional, controlled study is aimed to evaluate the efficacy and safety of cyclophosphamide in the treatment of idiopathic retroperitoneal fibrosis, which refers to the chronic nonspecific inflammation of retroperitoneal fascia and adipose tissue that gradually evolves into fibroproliferative disease.

DETAILED DESCRIPTION:
Idiopathic retroperitoneal fibrosis is a chronic disease that requires treatment for a few years. Patients with this disease respond well to glucocorticoid therapy, so you need to take glucocorticoid medication once the diagnosis is established. In addition, most patients need to use immunosuppressants when taking glucocorticoids. At present, the most commonly used immunosuppressants in the world are cyclophosphamide, azathioprine, methotrexate and mycophoranate, etc. The function of the above drugs is to improve the disorder of the immune system function, in order to restore the normal immune state, so that the inflammation and swelling of the affected organs disappear, restore the normal function. It should be emphasized that if the use of hormones and immunosuppressant is not standard or stopped too early, it can lead to disease recurrence. Therefore, after the disease is under control, long-term adherence to medication is needed to maintain a stable state of the disease.

At present, there is no clear treatment guideline for idiopathic retroperitoneal fibrosis in the world, and the addition of immunosuppressant is also out of debate. Therefore, a comprehensive evaluation of its pathogenesis, clinical characteristics and treatment response is needed.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 diagnosed as IRPF. The diagnosis of idiopathic retroperitoneal fibrosis is based on the following aspects :(1) the swelling of retroperitoneal tissue , which seems neoplastic; (2) A large number of lymphocytes proliferated and infiltrated in the affected tissues and organs, and tissues showed inflammation, fibrosis and sclerosis, in which IgG4-positive cells accounted for less than 50% of plasma cells; (3) Increased inflammatory markers, such as ESR and CRP; (4) Good response to glucocorticoid therapy.

Exclusion Criteria:

* malignancy retroperitoneal fibrosis secondary to other diseases or drugs or abdominal surgeries.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
remission | 5 years
  Patients achieve remission in symptoms and laboratory tets or radiologic images and have a low diseae activity after treatment.

SECONDARY OUTCOMES:
relapse | 5 years
  Patients have a recurrence of symptoms or laboratory abnormalities and have a considerable diseae activity after achieving remission.

OTHER OUTCOMES:
adverse events | 5 years
  Patients have adverse events due to the drug treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marzano A, Trapani A, Leone N, Actis GC, Rizzetto M. Treatment of idiopathic retroperitoneal fibrosis using cyclosporin. Ann Rheum Dis. 2001 Apr;60(4):427-8. doi: 10.1136/ard.60.4.427. PMID 11247880
- [Background] Vaglio A, Salvarani C, Buzio C. Retroperitoneal fibrosis. Lancet. 2006 Jan 21;367(9506):241-51. doi: 10.1016/S0140-6736(06)68035-5. PMID 16427494
- [Background] Jagadesham VP, Scott DJ, Carding SR. Abdominal aortic aneurysms: an autoimmune disease? Trends Mol Med. 2008 Dec;14(12):522-9. doi: 10.1016/j.molmed.2008.09.008. Epub 2008 Nov 6. PMID 18980864
- [Background] Qian Q, Kashani KB, Miller DV. Ruptured abdominal aortic aneurysm related to IgG4 periaortitis. N Engl J Med. 2009 Sep 10;361(11):1121-3. doi: 10.1056/NEJMc0905265. No abstract available. PMID 19741239
- [Background] Scheel PJ Jr, Feeley N, Sozio SM. Combined prednisone and mycophenolate mofetil treatment for retroperitoneal fibrosis: a case series. Ann Intern Med. 2011 Jan 4;154(1):31-6. doi: 10.7326/0003-4819-154-1-201101040-00005. PMID 21200036
- [Background] Vaglio A, Palmisano A, Alberici F, Maggiore U, Ferretti S, Cobelli R, Ferrozzi F, Corradi D, Salvarani C, Buzio C. Prednisone versus tamoxifen in patients with idiopathic retroperitoneal fibrosis: an open-label randomised controlled trial. Lancet. 2011 Jul 23;378(9788):338-46. doi: 10.1016/S0140-6736(11)60934-3. Epub 2011 Jul 4. PMID 21733570
- [Background] Binder M, Uhl M, Wiech T, Kollert F, Thiel J, Sass JO, Walker UA, Peter HH, Warnatz K. Cyclophosphamide is a highly effective and safe induction therapy in chronic periaortitis: a long-term follow-up of 35 patients with chronic periaortitis. Ann Rheum Dis. 2012 Feb;71(2):311-2. doi: 10.1136/annrheumdis-2011-200148. Epub 2011 Aug 22. No abstract available. PMID 21859695
- [Background] Alberici F, Palmisano A, Urban ML, Maritati F, Oliva E, Manenti L, Ferretti S, Cobelli R, Buzio C, Vaglio A. Methotrexate plus prednisone in patients with relapsing idiopathic retroperitoneal fibrosis. Ann Rheum Dis. 2013 Sep 1;72(9):1584-6. doi: 10.1136/annrheumdis-2013-203267. Epub 2013 May 21. No abstract available. PMID 23696631
- [Background] Fatima J, Gota C, Clair DG, Billings SD, Gornik HL. Inflammatory abdominal aortic aneurysm with retroperitoneal fibrosis. Circulation. 2014 Oct 7;130(15):1300-2. doi: 10.1161/CIRCULATIONAHA.114.010173. No abstract available. PMID 25287771
- [Background] Fernando A, Pattison J, Horsfield C, D'Cruz D, Cook G, O'Brien T. [18F]-Fluorodeoxyglucose Positron Emission Tomography in the Diagnosis, Treatment Stratification, and Monitoring of Patients with Retroperitoneal Fibrosis: A Prospective Clinical Study. Eur Urol. 2017 Jun;71(6):926-933. doi: 10.1016/j.eururo.2016.10.046. Epub 2016 Nov 18. PMID 27876167